CLINICAL TRIAL: NCT03593174
Title: Étude de l'efficacité du Pansement Rigide Amovible Sous Vide à Titre de modalité de Pansement Post-amputation Tibiale
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-2617
Record Dates: First submitted 2018-06-19; First posted 2018-07-19 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Trans-tibial Amputations
Keywords: Amputation
MeSH Terms: interventions — Compression Bandages

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ossur Rigid Dressing (Experimental): Use of ORD, which is a type of Removable Rigid Dressing (RRD), as a post tibial amputation dressing modality.
  Interventions: Device: Ossur Rigid Dressing
- Elastic bandage (Active Comparator): Use of the elastic bandage as a post amputation dressing modality.
  Interventions: Device: Elastic Bandage

INTERVENTIONS:
Device: Ossur Rigid Dressing — Removable Rigid Dressing
  Arms: Ossur Rigid Dressing
Device: Elastic Bandage — Usual modality: Elastic bandage
  Arms: Elastic bandage

SUMMARY:
The present study will measure the efficiency of a new modality for trans-tibial amputations in Quebec's health system, to reduce the time before prosthesis fitting, compared to the usual modality. The present study will evaluate the feasability of implantation of this new modality in Quebec and demonstrate its superiority in comparison to the usual modality (shorter time before fitting and reduction of costs).

DETAILED DESCRIPTION:
The main objective of the present study is to obtain an estimation of the efficiency of a Removable Rigid Dressing (RRD) -type compression modality immediately following a tibial amputation as an alternative to the elastic bandage, which is the usually-used modality. This pilot study will verify the feasability of implantation of this type of dressing, and to collect data on the main dependant variables of this research projet in order to eventually estimate the expected effect on a larger population.

The main objectives of this study are:

1. To explore the efficacy of the RRD in comparison to the elastic bandage on the size of the stump, associated complications and necessary time to fitting of the prosthesis.
2. Verify the facilitators and obstacles to implantation of the RRD as a post tibial ambutation dressing modality as an alternative to the elastic bandage.

ELIGIBILITY:
Inclusion Criteria:

* Need of a trans-tibial amputation of atraumatic cause
* Between 40 and 75 years of age

Exclusion Criteria:

- Having a medical condition that could significantly affect the healing process

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Stump size | 8 weeks
  Leg circumference measure

CONTACTS AND LOCATIONS:
Overall Officials: Michel Tousignant, Phd, Study Director — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No